CLINICAL TRIAL: NCT02560727
Title: Feasibility, Safety, and Efficacy of Transendoscopic Enteral Tubing in Fecal Microbiota Transplantation
Brief Title: To Evaluate the Feasibility, Safety, and Efficacy of TET for FMT Via Colonic Approach
Acronym: TET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Collaborators: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Faming Zhang, Associate professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Other Study IDs: TET-CN-121002
Record Dates: First submitted 2015-09-21; First posted 2015-09-25 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Inflammatory Bowel Diseases; Fecal Microbiota Transplantation; transendoscopic enteral tubing
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Colonoscopes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- colonoscope via of FMT: FMT pathway is colonoscope
  Interventions: Device: colonoscope
- Transendoscopic enteral tubing: FMT was performed via TET tube
  Interventions: Device: transendoscopic enteral tubing

INTERVENTIONS:
Device: transendoscopic enteral tubing — Investigators designed transendoscopic enteral tubing (TET).The enteral segment of the tube is fixed in the ileocecum with distal segment fixed buttocks. The tube was used for FMT and colonic local administration
  Other Names: TET
  Groups: Transendoscopic enteral tubing
Device: colonoscope — FMT via colonoscope is the most common approach.
  Groups: colonoscope via of FMT

SUMMARY:
No technique by placing a tube through anus into cecum for whole colon administration. This study aimed to evaluate the feasibility, safety, and efficacy of transendoscopic enteral tubing (TET) in fecal microbiota transplantation (FMT) through whole colon.

DETAILED DESCRIPTION:
The previous reported fecal microbiota transplantation (FMT)through whole colon. delivering ways were involved with upper digestive tract, middle digestive tract and lower digestive tract. FMT via colonoscope is the most common approach, participants have to endure the discomfortable of bowel preparation and colonoscopy, and FMT by colonoscopy was recommended for repeat FMT treatment in short period. Traditional enema infuses bacteria solution into rectal and sigmoid colon but cannot spread to whole colon.No technique by placing a tube through anus into cecum for whole colon administration, which could be maintained for repeat FMTs.To solve these problems, investigators designed a new technique called transendoscopic enteral tubing (TET).the TET tube was fixed at cecum by clips under endoscopy. This study aimed to evaluate the feasibility, safety, and efficacy of TET for FMT via colonic approach.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate ulcerative colitis (Montreal classification)

Exclusion Criteria:

* Diagnosed as ulcerative colitis first time.
* No history of using Biologic, immunomodulatory therapy or corticosteroid therapy.
* With contraindication of endoscopy.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A prospective study was conducted at the Digestive Medicine Center of the Second Affiliated Hospital of Nanjing Medical University from October 2014 to June 2016. All recruited cases met the including criteria: aged 10-70 yr, suitable for endoscopy, and agreed to undergo FMT and TET
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
durability of clinical remission | One year
  The durability of clinical remission (days) after Fecal Microbiota Transplantation procedure by TET.Defined as Montreal score S0 (clinical remission)

SECONDARY OUTCOMES:
Patients with worsened disease | one year
  Number of patients with worsened disease. Increase in Montreal score S1, S2 and S3.

OTHER OUTCOMES:
Adverse events | one year
  Number of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, MD,PhD, Principal Investigator — Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University
Locations (1):
- Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Youngster I, Russell GH, Pindar C, Ziv-Baran T, Sauk J, Hohmann EL. Oral, capsulized, frozen fecal microbiota transplantation for relapsing Clostridium difficile infection. JAMA. 2014 Nov 5;312(17):1772-8. doi: 10.1001/jama.2014.13875. PMID 25322359
- [Background] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Background] Cui B, Feng Q, Wang H, Wang M, Peng Z, Li P, Huang G, Liu Z, Wu P, Fan Z, Ji G, Wang X, Wu K, Fan D, Zhang F. Fecal microbiota transplantation through mid-gut for refractory Crohn's disease: safety, feasibility, and efficacy trial results. J Gastroenterol Hepatol. 2015 Jan;30(1):51-8. doi: 10.1111/jgh.12727. PMID 25168749
- [Derived] Ding X, Li Q, Li P, Zhang T, Cui B, Ji G, Lu X, Zhang F. Long-Term Safety and Efficacy of Fecal Microbiota Transplant in Active Ulcerative Colitis. Drug Saf. 2019 Jul;42(7):869-880. doi: 10.1007/s40264-019-00809-2. PMID 30972640